CLINICAL TRIAL: NCT04801550
Title: Study of Somatosensory Responses During Millimeter Waves Application (RESOM)
Brief Title: Study of Somatosensory Responses During Millimeter Waves Application
Acronym: RESOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government); Remedee SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 38RC20.370
Record Dates: First submitted 2021-03-05; First posted 2021-03-17 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers
Keywords: Somatosensory stimulus; Millimeter Waves; Magnetoencephalography

STUDY DESIGN:
Intervention Model Description: This is an exploratory and prospective study. Each volunteer will undergo two MEG examinations (4h-long each) without knowing the millimeter wave emitter status. Each volunteer acts as their own control. The status of exposure to millimeter waves is randomized.
  The study is cross-over and double-blinded.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Millimeter wave emitter status 1 (Active Comparator): Somatosensory stimulus during Magnetoencephalography (MEG) records
  Interventions: Device: Millimeter waves local exposure
- Millimeter wave emitter status 2 (Sham Comparator): Somatosensory stimulus during Magnetoencephalography (MEG) records
  Interventions: Device: Millimeter waves local exposure

INTERVENTIONS:
Device: Millimeter waves local exposure — several blocks of somatosensory evoked potentials with or without Millimeter waves local exposure

SUMMARY:
The brain activity induced by a sensory stimulus and measured by magnetoencephalography will be compared before and after exposure to millimeter waves. We hypothesize that brain activity is modified after exposure to millimeter waves. The neuromodulatory effects of millimeter waves may lead to future development on therapeutic management in anxiety and pain.

DETAILED DESCRIPTION:
Several studies showed clinical efficacy of millimeter waves in pain management, with no side-effects.

However, its mechanism of action is still partly unknown. Preclinical studies showed that the use of millimeter waves near highly-innervated areas stimulates subcutaneous receptors, even at low power.

To achieve safe millimeter wave stimulation, we will use a bracelet (Remedee Labs) emitting millimeter waves, that has been developped for human use. It complies with radiofrequency exposure regulation (CE-marked).

This study aims to provide a better understanding of the mechanism by which millimeter waves interact with somatosensory system in brain.

For this purpose, the analysis of brain activity will focus on somatosensory responses elicited by electrical stimulation of the right thumb.

Subjects will complete two sessions during which the brain activity will be recorded by magnetoencephalography (MEG) before, during and after the use of a bracelet emitting millimeter waves.

Magnetoencephalography is chosen for its good temporal resolution, its sensitivity in the low frequencies and its accuracy to locate neural sources when matching with an Magnetic Resonance (MR) Imagery. It will allow us to study the shape and the delay of the somatosensory response in primary somatosensory cortex (SI) and secondary somatosensory cortex (SII) cortical areas of the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male voluntary subject, aged 18 to 40 inclusive.
2. Right-handed subject verified by the Edinburgh test.
3. Body mass index (BMI) between 18 and 25 kg/m2 inclusive.
4. Blood pressure and heart rate considered clinically normal by the investigators.
5. Having benefited from a medical examination before participating in the research.
6. Volunteer with a wrist circumference between 14.5 and 21 cm (wrist compatible with the size of the bracelet).
7. Adults, having expressed their consent to research, affiliated to a social security scheme and registered in the national file of people who lend themselves to biomedical research

Exclusion Criteria:

1. Any history or presence of chronic disease.
2. Volunteer presenting chronic pain and / or headache.
3. Metal or silicon allergy.
4. Volunteer with a piercing or an implanted metallic material on the internal face of the right wrist.
5. Volunteer with a tattoo on the inside of the right wrist.
6. People with contraindications to MRI.
7. Taking treatment that could impact the physiological measurements recorded.
8. Consumption of analgesics or anti-inflammatory drugs during the week before each MEG examination.
9. Surgical intervention within the last 3 months.
10. Alcohol consumption within the last 24 hours, for each visit.
11. Achievement of a sporting effort within the last 24 hours, for each visit.
12. Volunteer with difficulties to be cooperative during the study in the opinion of the investigator (i.e.: language problem, poor mental development, etc.).
13. Volunteer in period of exclusion from another study.
14. Volunteer deprived of liberty by a judicial or administrative decision, subject to psychiatric treatment, or major subject subject to a legal protection measure (guardianship, guardianship and safeguard of justice) referred to in articles 1121-6 to 1121-8 of the French public health code.
15. Volunteer who would receive more than 4,500 euros in compensation as a result of his participation in other research involving the human person in the 12 months preceding this study.
16. Volunteer who cannot be contacted in case of emergency.
17. Volunteer who have already used an millimeter wave emitter before the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Change in the somatosensory responses induced by the application of millimeter waves to the wrist | 4 hours
  Statistically significant change in the evoked somatosensory magnetic activity time course

SECONDARY OUTCOMES:
Variation of the sympathovagal balance following the application of millimeter waves | 4 hours
  Comparison of heart rate variability before and after application of millimeter waves
Changes in resting brain activity during or after application of millimeter waves to the wrist | 4 hours
  Characterization of oscillatory brain activity by frequency bands (power maps)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinatec Cea/Chuga, Grenoble, France

REFERENCES:
- [Background] Fioravanti C, Kajal SD, Carboni M, Mazzetti C, Ziemann U, Braun C. Inhibition in the somatosensory system: An integrative neuropharmacological and neuroimaging approach. Neuroimage. 2019 Nov 15;202:116139. doi: 10.1016/j.neuroimage.2019.116139. Epub 2019 Aug 30. PMID 31476429
- [Background] Radzievsky AA, Gordiienko OV, Alekseev S, Szabo I, Cowan A, Ziskin MC. Electromagnetic millimeter wave induced hypoalgesia: frequency dependence and involvement of endogenous opioids. Bioelectromagnetics. 2008 May;29(4):284-95. doi: 10.1002/bem.20389. PMID 18064600
- [Background] Rojavin MA, Ziskin MC. Electromagnetic millimeter waves increase the duration of anaesthesia caused by ketamine and chloral hydrate in mice. Int J Radiat Biol. 1997 Oct;72(4):475-80. doi: 10.1080/095530097143248. PMID 9343112